CLINICAL TRIAL: NCT06081153
Title: A Randomized, Placebo-Controlled Mechanistic Clinical Trial of PCSK9 Inhibition With Evolocumab in Patients Undergoing Open Abdominal Aortic Aneurysm Repair
Brief Title: Mechanistic Clinical Trial of PCSK9 Inhibition for AAA
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Amgen (Industry)
Responsible Party: Principal Investigator, Scott Damrauer, Associate Professor of Surgery, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 852428; R01HL166991 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Evolocumab (Experimental): Evolocumab is the drug that will be administered in this study. It will be administered as a 140mg subcutaneous injection every 14 days for 5 weeks (for a total of 3 doses).
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): This arm is a matching placebo that will be administered in the same fashion as the study drug if the patient is randomized to placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab — See arm description.
  Arms: Evolocumab
Drug: Placebo — See arm description.
  Arms: Placebo

SUMMARY:
The goal of this mechanistic clinical trial is to assess whether lowering the low-density lipoprotein cholesterol (LDL-C) levels in the blood with the injections of the medication evolocumab will have any effect on the tissue or cells of patients with abdominal aortic aneurysm (AAA). Researchers will compare participants receiving evolocumab injections to participants receiving placebo injections to see how the tissue and cells of the aorta are affected by changes in LDL-C levels.

DETAILED DESCRIPTION:
After being informed about the study and its potential risks, all patients giving informed consent will undergo a baseline visit and be randomized to received either evolocumab 140mg subcutaneously or placebo. This baseline visit includes a vital signs assessment, laboratory tests, medical history and medication review, a pregnancy test (if applicable), and training on how to perform drug injections. Participants will receive 3 doses/autoinjectors of study drug or placebo and be instructed to perform injections every 14 days starting 5 weeks prior to their scheduled AAA repair. If the baseline assessment occurs 5 weeks prior to their scheduled AAA, the first injection will be performed during this visit. Participants will have the option of coming back to the site for injections 2 and 3 or perform these injections at home under telehealth supervision. At the time of open AAA repair, participants will repeat laboratory tests and have a sample of aneurysm tissue taken. Participants will then have a follow up phone call 4 weeks after AAA repair to assess for any adverse events. At the conclusion of the study investigators will examine gene expression and protein levels in the aortic tissue to determine the impact of LDL-C lowering with evolocumab.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal aortic aneurysm (AAA) requiring open surgical repair
2. Age > 18
3. Provision of signed and dated informed consent form
4. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Prior use of a PCSK9 inhibitor (evolocumab, alirocumab, inclisiran) within 6 months of the baseline visit
2. LDL-C < 40 mg/dL (within 3 months of baseline visit)
3. Known allergy to PCSK9 inhibitor
4. Aortic dissection
5. Vascular connective tissue disorders
6. Type I-III or V Thoraco-abdominal Aortic Aneurysm
7. Vasculitis or inflammatory aneurysm
8. Pregnant or lactating women
9. Poorly controlled diabetes (A1C > 10%)
10. Chronic kidney disease Stage 4/5 or End Stage Renal Disease (ESRD) on hemodialysis (HD)
11. Liver Disease (alanine transaminase [ALT] or aspartate aminotransferase [ALT] > 3.0 x upper limits of normal) (within 3 months of baseline visit)
12. Known latex or naturally rubber allergy
13. Treatment with another investigational product within 30 days or 5 half-lives of the investigation drug before consent (whichever is longer) that would have an impact on endpoints associated with this trial.
14. Any other condition that the Investigator feels prohibits participants' ability to comply with study or follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Interleukin (IL)-6 in myeloid derived monocytes/macrophages from in AAA tissue | AAA Repair (Week 5)
  IL-6 expression will be measured in myeloid cells in the aortic tissue specimens using single nucleus RNA sequencing and confirmed by whole tissue ELISA.

SECONDARY OUTCOMES:
Matrix metalloproteinase (MMP)-9 in myeloid derived monocytes/macrophages from in AAA tissue | AAA Repair (Week 5)
  MMP-9 expression will be measured in myeloid cells in the aortic tissue specimens using single nucleus RNA sequencing and confirmed by whole tissue ELISA and immunofluorescence activity assays.
Infiltrating immune cell composition and their activation/inflammatory states in AAA tissue | AAA Repair (Week 5)
  Relative numbers of infiltrating immune cell type and their activation/inflammatory state as measured by a combination of bulk and single nuclear RNA sequencing
Smooth muscle composition of AAA tissue | AAA Repair (Week 5)
  The relative numbers of smooth muscle cells and their contractile/proliferative state as measured by a combination of bulk and single nucleus RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Scott Damrauer, MD, Principal Investigator — University of Pennsylvania